CLINICAL TRIAL: NCT02947516
Title: Comparison of Pain Scores Between Endoscopic Ultrasound (EUS)-Guided Liver Biopsy and Percutaneous Liver Biopsy
Brief Title: Comparison of EUS-Guided Liver Biopsy With Percutaneous Liver Biopsy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding n/a
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Marvin Ryou, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 20162017
Record Dates: First submitted 2016-10-25; First posted 2016-10-28 (Estimated); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Fibrosis
Keywords: Endoscopic Ultrasound-Guided Fine Needle Aspiration; liver; biopsy; pain
MeSH Terms: conditions — Fibrosis; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Percutaneous liver biopsy (Active Comparator): Participants will be referred for liver biopsy by their hepatologist/gastroenterologist. The intervention is that these participants will undergo a percutaneous liver biopsy per standard protocol.
  Interventions: Procedure: Percutaneous liver biopsy
- EUS-guided liver biopsy (Experimental): Participants will be referred for liver biopsy by their hepatologist/gastroenterologist. The intervention is that these participants will undergo an endoscopic ultrasound procedure per standard protocol. The liver will be identified, and Color Doppler imaging prior to needle puncture will confirm lack of significant vascular structures within the needle path. Liver biopsies using up to 1-2 passes from the left hepatic lobe using a transgastric approach and up to 1-2 passes from the right hepatic lobe using a transduodenal bulb approach will be performed. The participant will be observed in the recovery unit for up to 60 minutes after the EUS-LB, and discharged if no pain or signs of complication.
  Interventions: Procedure: Endoscopic ultrasound-guided liver biopsy

INTERVENTIONS:
Procedure: Endoscopic ultrasound-guided liver biopsy — Participants will undergo endoscopic ultrasound per standard technique, with liver biopsy performed at that time.
  Arms: EUS-guided liver biopsy
Procedure: Percutaneous liver biopsy — Participants will undergo percutaneous liver biopsy per standard protocol.
  Arms: Percutaneous liver biopsy

SUMMARY:
There are several ways to perform liver biopsies, including the percutaneous route (historical gold standard) and via endoscopic ultrasound (EUS) guidance. The primary aim of this study is to prospectively compare patients undergoing EUS-guided liver biopsies to patients undergoing percutaneous biopsy. The investigators hypothesize that (1) patients who are randomized to undergo EUS-guided liver biopsy will rate themselves as having less pain in the 48 hours following the procedure, and (2) will have comparable histologic yield to a 2:1 matched cohort of patients undergoing percutaneous liver biopsies.

DETAILED DESCRIPTION:
Currently, liver biopsy is the gold standard for determining the index of liver fibrosis in a patient with chronic liver disease, and whether the patient has progressed to cirrhosis. These biopsies are predominantly performed percutaneously. However, there are several complications related to liver biopsy, the most common of which are pain and bleeding.

There has been significant movement over the past several years to assess the utility of alternative techniques and approaches for the evaluation of liver disease. Endoscopic ultrasound (EUS) is a well-established technique for diagnostic and therapeutic evaluation of gastrointestinal and pancreaticobiliary disorders. EUS-guided liver biopsy (EUS-LB) has shown to be technically simple, safe, and provides adequate diagnostic yield for evaluation of liver disease in both children and adults. There are several advantages to EUS-LB. First, it would theoretically be less painful than the percutaneous approach, as it does not require skin puncture and also offers the comfort of sedation and analgesia. It also eliminates the need for breath hold. Furthermore, it is an image-guided approach which allows visualization and avoidance of blood vessels even 1 mm in size. Additionally, it provides an access area to a much wider segment of liver parenchyma as the entire left lobe, and the majority of the right lobe can be evaluated for possible needle puncture sites from the stomach and duodenal bulb, respectively. In addition to obtaining tissue, EUS-LB also offers the benefit of evaluating the biliary tree, gallbladder, pancreas, lymph nodes, and vascular anatomy for a more comprehensive evaluation in the same setting. Finally, in patients ultimately found to have biopsy-proven cirrhosis, it simultaneously provides the necessary variceal screening which would otherwise require an additional procedure.

The aim of this study is to prospectively perform EUS-guided liver biopsies in patients who are otherwise candidates for percutaneous biopsy. We hypothesize that (1) patients who are randomized to undergo EUS-guided liver biopsy will rate themselves as having less pain in the 48 hours following the procedure and (2) will have comparable histologic yield to a 2:1 matched cohort of patients undergoing percutaneous transjugular liver biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Eligibility for receiving conscious sedation or monitored anesthesia care
* Abnormal liver function tests with comprehensive previous evaluation (including serologic testing and cross-sectional imaging) leading to an appropriate decision to proceed with liver biopsy and/or portal pressure measurements.

Exclusion Criteria:

* Suspected or known malignant liver disease
* Severe thrombocytopenia (platelets <50,000/microL)
* Severe coagulopathy (international normalized ratio [INR] > 1.7 or other known coagulopathy)
* Use of antiplatelet agents within 7 days of the procedure
* Inability to provide informed consent
* Pregnancy or suspected pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Pain Scores on the Universal Pain Assessment Tool (UPAT) | 48 hours

SECONDARY OUTCOMES:
Pain Medication Requirements | 48 hours
  Use of any analgesics/narcotics
Histologic Yield | 1 week
  Number of portal triads on histology

CONTACTS AND LOCATIONS:
Overall Officials: Marvin Ryou, MD, Principal Investigator — Brigham and Women's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bedossa P, Dargere D, Paradis V. Sampling variability of liver fibrosis in chronic hepatitis C. Hepatology. 2003 Dec;38(6):1449-57. doi: 10.1016/j.hep.2003.09.022. PMID 14647056
- [Result] Eisenberg E, Konopniki M, Veitsman E, Kramskay R, Gaitini D, Baruch Y. Prevalence and characteristics of pain induced by percutaneous liver biopsy. Anesth Analg. 2003 May;96(5):1392-1396. doi: 10.1213/01.ANE.0000060453.74744.17. PMID 12707140
- [Result] Caldwell SH. Controlling pain in liver biopsy, or "we will probably need to repeat the biopsy in a year or two to assess the response". Am J Gastroenterol. 2001 May;96(5):1327-9. doi: 10.1111/j.1572-0241.2001.03847.x. No abstract available. PMID 11374664
- [Result] Piccinino F, Sagnelli E, Pasquale G, Giusti G. Complications following percutaneous liver biopsy. A multicentre retrospective study on 68,276 biopsies. J Hepatol. 1986;2(2):165-73. doi: 10.1016/s0168-8278(86)80075-7. PMID 3958472
- [Result] Huang JF, Hsieh MY, Dai CY, Hou NJ, Lee LP, Lin ZY, Chen SC, Wang LY, Hsieh MY, Chang WY, Yu ML, Chuang WL. The incidence and risks of liver biopsy in non-cirrhotic patients: An evaluation of 3806 biopsies. Gut. 2007 May;56(5):736-7. doi: 10.1136/gut.2006.115410. No abstract available. PMID 17440193
- [Result] Perrault J, McGill DB, Ott BJ, Taylor WF. Liver biopsy: complications in 1000 inpatients and outpatients. Gastroenterology. 1978 Jan;74(1):103-6. PMID 618417
- [Result] Firpi RJ, Soldevila-Pico C, Abdelmalek MF, Morelli G, Judah J, Nelson DR. Short recovery time after percutaneous liver biopsy: should we change our current practices? Clin Gastroenterol Hepatol. 2005 Sep;3(9):926-9. doi: 10.1016/s1542-3565(05)00294-6. PMID 16234032
- [Result] Stone MA, Mayberry JF. An audit of ultrasound guided liver biopsies: a need for evidence-based practice. Hepatogastroenterology. 1996 Mar-Apr;43(8):432-4. PMID 8714240
- [Result] Hollerbach S, Willert J, Topalidis T, Reiser M, Schmiegel W. Endoscopic ultrasound-guided fine-needle aspiration biopsy of liver lesions: histological and cytological assessment. Endoscopy. 2003 Sep;35(9):743-9. doi: 10.1055/s-2003-41593. PMID 12929021
- [Result] Fuccio L, Larghi A. Endoscopic ultrasound-guided fine needle aspiration: How to obtain a core biopsy? Endosc Ultrasound. 2014 Apr;3(2):71-81. doi: 10.4103/2303-9027.123011. PMID 24955336
- [Result] Stavropoulos SN, Im GY, Jlayer Z, Harris MD, Pitea TC, Turi GK, Malet PF, Friedel DM, Grendell JH. High yield of same-session EUS-guided liver biopsy by 19-gauge FNA needle in patients undergoing EUS to exclude biliary obstruction. Gastrointest Endosc. 2012 Feb;75(2):310-8. doi: 10.1016/j.gie.2011.09.043. PMID 22248599
- [Result] Iglesias-Garcia J, Poley JW, Larghi A, Giovannini M, Petrone MC, Abdulkader I, Monges G, Costamagna G, Arcidiacono P, Biermann K, Rindi G, Bories E, Dogloni C, Bruno M, Dominguez-Munoz JE. Feasibility and yield of a new EUS histology needle: results from a multicenter, pooled, cohort study. Gastrointest Endosc. 2011 Jun;73(6):1189-96. doi: 10.1016/j.gie.2011.01.053. Epub 2011 Mar 21. PMID 21420083
- [Result] Johal AS, Khara HS, Maksimak MG, Diehl DL. Endoscopic ultrasound-guided liver biopsy in pediatric patients. Endosc Ultrasound. 2014 Jul;3(3):191-4. doi: 10.4103/2303-9027.138794. PMID 25184126